CLINICAL TRIAL: NCT00327184
Title: Study to Demonstrate Non-inferiority of GSK Biologicals' Hib-MenC Given With Infanrix™ Penta Versus NeisVac-C™ Given With Infanrix™ Hexa at 3, 5 Months of Age and Persistence Prior to a Hib-MenC Booster at 11 Months and Immunogenicity of the Booster
Brief Title: Primary & Booster Study in Infants to Demonstrate Non-inferiority, Persistence & Immunogenicity of Hib-MenC Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 106388; 106390 (Other: GSK)
Record Dates: First submitted 2006-05-16; First posted 2006-05-18 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-10

CONDITIONS: Neisseria Meningitidis; Haemophilus Influenzae Type b
MeSH Terms: conditions — Haemophilus Infections | interventions — Vaccines; diphtheria-tetanus-acellular pertussis-inactivated poliovirus-Haemophilus influenzae b conjugate-hepatitis B vaccine

ARMS (2):
- Group Hib-MenC (Experimental): Subjects receive 2 primary vaccination doses at 3 and 5 months of age and a booster dose at 11 months of age of Hib-MenC + Infanrix™ penta vaccines.
  Interventions: Biological: Haemophilus influenzae type b- and meningococcal serogroup C (vaccine); Biological: Infanrix Penta
- Group NeisVac-C (Active Comparator): Subjects receive 2 primary vaccination doses at 3 and 5 months of age and a booster dose at 11 months of age of NeisVac-C™ + Infanrix™ hexa vaccines.
  Interventions: Biological: Infanrix hexa; Biological: Neis-Vac-C

INTERVENTIONS:
Biological: Haemophilus influenzae type b- and meningococcal serogroup C (vaccine) — Two primary vaccination doses at 3 and 5 months of age and a booster dose at 11 months of age.
  Arms: Group Hib-MenC
Biological: Infanrix Penta — Two primary vaccination doses at 3 and 5 months of age and a booster dose at 11 months of age.
  Arms: Group Hib-MenC
Biological: Infanrix hexa — Two primary vaccination doses at 3 and 5 months of age and a booster dose at 11 months of age
  Arms: Group NeisVac-C
Biological: Neis-Vac-C — Two primary vaccination doses at 3 and 5 months of age and a booster dose at 11 months of age
  Arms: Group NeisVac-C

SUMMARY:
The purpose of this primary vaccination phase is to demonstrate the non-inferiority of two doses of Biologicals' Hib-MenC conjugate vaccine when given with Infanrix™ penta to infants (at 3 & 5m) compared to NeisVac-C™ given with Infanrix™ hexa.

The purpose of the booster vaccination phase is to evaluate the immunogenicity, safety and reactogenicity of a booster dose of the Hib-MenC vaccine given with Infanrix™ penta at 11 m of age versus NeisVac-C™ given with Infanrix™ hexa, as well as the antibody persistence prior to the administration of the booster doses. The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

DETAILED DESCRIPTION:
This multicenter study is open and consists of a primary and a booster phase. The study has 2 treatment groups with NeisVac-C™ + Infanrix™ hexa as active controls. In the primary phase, one blood sample will be collected from all subjects for immunogenicity analyses- one month after the second vaccination dose. In the booster phase, two blood samples will be collected: prior to and one month post booster vaccination.

ELIGIBILITY:
Inclusion Criteria

Primary Phase:

* Subjects who the investigator believes that their parents/guardians can and will comply with the requirements of the protocol should be enrolled in the study.
* healthy male or female subject between, and including, 6 and 12 weeks of age at the time of the first vaccination, born after a gestation period between and including 36 and 42 weeks.
* Written informed consent obtained from the parent or guardian of the subject prior to the study entry.
* Free of obvious health problems as established by medical history and clinical examination before entering into the study.

Booster Phase:

• Participation in primary phase of study.

Exclusion Criteria

Primary Phase:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) since birth or planned use during the study period.
* Chronic administration (defined as more than 14 days) of immunosuppressant or other immune-modifying drugs since birth.
* Planned administration/ administration of a vaccine not foreseen by the study protocol since birth, with exception of BCG.
* Previous vaccination against meningococcal serogroup C disease, diphtheria, tetanus, pertussis, polio, pneumococcal, Hepatitis B or Hib disease
* History of Haemophilus influenzae type b and /or meningococcal serogroup C disease.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus infection.
* A family history of congenital or hereditary immunodeficiency.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Major congenital defects or serious chronic illness.
* History of any neurologic disorders or seizures.
* Acute disease at the time of enrolment.
* Administration of immunoglobulins and/or any blood products since birth or planned administration during the study period.

Additional Exclusion criteria for the Booster Phase:

• Previous booster vaccination with Hib and/or MenC and/or DTP containing and/or IPV containing and/or HepB containing vaccine(s).

Ages: 6 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 709 (Actual)
Dates: Start 2006-04; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
SBA-MenC titre | One month after the second dose of the Primary Vaccination Phase.
Anti-PRP concentration | One month after the second dose of the Primary Vaccination Phase

SECONDARY OUTCOMES:
SBA-MenC titres | One month after the second dose of the Primary Vaccination Phase; prior to and one month after the Booster Vaccination
Anti-PRP concentrations | One month after the second dose of the Primary Vaccination Phase; prior to and one month after the Booster Vaccination
Anti-PSC concentrations | One month after the second dose of the Primary Vaccination Phase; prior to and one month after the Booster Vaccination.
Anti-HBs concentrations | One month after the second dose of the Primary Vaccination Phase; prior to and one month after the Booster Vaccination
Occurrence of local solicited adverse events. | During the solicited follow-up period (Day 0 - Day 3) following the administration of each vaccine dose.
Occurrence of solicited general adverse events | During the solicited follow-up period (Day 0 - Day 3) following the administration of each vaccine dose.
Occurrence of unsolicited non-serious adverse events | Within 30 days after each vaccination
Occurrence of any serious adverse events | Throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (14):
- Finland (10):
  - GSK Investigational Site, Espoo
  - GSK Investigational Site, Helsinki
  - GSK Investigational Site, Jarvenpaa
  - GSK Investigational Site, Kotka
  - GSK Investigational Site, Lahti
  - GSK Investigational Site, Oulu
  - GSK Investigational Site, Pori
  - GSK Investigational Site, Tampere
  - GSK Investigational Site, Turku
  - GSK Investigational Site, Vantaa
- Italy (4):
  - GSK Investigational Site, Bari, Apulia
  - GSK Investigational Site, Lodi, Lombardy
  - GSK Investigational Site, Sassari, Sardinia
  - GSK Investigational Site, Ragusa, Sicily

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Vesikari T, Forsten A, Desole MG, Ferrera G, Caubet M, Mesaros N, Boutriau D. A combined Haemophilus influenzae type B Neisseria meningitidis serogroup C tetanus toxoid conjugate vaccine is immunogenic and well-tolerated when coadministered with diphtheria, tetanus, acellular pertussis hepatitis B-inactivated poliovirus at 3, 5 and 11 months of age: results of an open, randomized, controlled study. Pediatr Infect Dis J. 2013 May;32(5):521-9. doi: 10.1097/INF.0b013e31827e22e3. PMID 23190785
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 106388 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 106388 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 106388 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 106388 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 106388 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 106388 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register. The results of this study 106388 are summarised with study 106390 on the GSK Clinical Study Register.